CLINICAL TRIAL: NCT00371683
Title: A Phase 3 Randomized, Double-Blind Active-Controlled (Enoxaparin), Parallel-Group, Multi-Center Study to Evaluate the Safety and Efficacy of Oral Apixaban in Subjects Undergoing Elective Total Knee Replacement Surgery
Brief Title: Study of Apixaban for the Prevention of Thrombosis-related Events Following Knee Replacement Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CV185-034
Record Dates: First submitted 2006-08-30; First posted 2006-09-04 (Estimated); Results first posted 2015-12-30 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-11

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism
Keywords: Prevention of deep vein thrombosis and pulmonary embolism after total knee replacement surgery
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — Enoxaparin; apixaban

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A1 (Active Comparator): + placebo
  Interventions: Drug: Enoxaparin + Placebo
- A2 (Experimental): + placebo
  Interventions: Drug: Apixaban + Placebo

INTERVENTIONS:
Drug: Enoxaparin + Placebo — Syringes + tablets, Subcutaneous + Oral, 30mg, twice daily, 12 day treatment period
  Other Names: Lovenox®
  Arms: A1
Drug: Apixaban + Placebo — Tablet + Syringes, Oral + subcutaneous, 2.5 mg, twice daily, 12 day treatment period
  Arms: A2

SUMMARY:
The purpose of this study is to learn if apixaban can prevent blood clots in the leg (deep vein Thrombosis [DVT]) and lung (pulmonary embolism [PE]) that sometimes occur after knee replacement surgery and to learn how apixaban compares to enoxaparin (Lovenox®) for preventing these clots. The safety of apixaban will also be studied.

ELIGIBILITY:
Key Inclusion Criteria:

* Men and non-pregnant, non-breastfeeding women
* 18 years or older
* Scheduled for knee replacement surgery

Key Exclusion Criteria:

* hereditary or acquired bleeding disorders
* clotting disorders
* bleeding or high risk for bleeding
* drugs that affect bleeding or coagulation
* need for ongoing parenteral or oral anticoagulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3608 (Actual)
Dates: Start 2006-11; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (96):
- United States (24):
  - Capstone Clinical Trials, Inc, Birmingham, Alabama
  - West Alabama Research, Inc., Tuscaloosa, Alabama
  - Martin Bowen Hefley Orthopedics, Little Rock, Arkansas
  - Colorado Orthopedic Consultants, Pc, Aurora, Colorado
  - Colorado Joint Replacement, Denver, Colorado
  - Jdpmedical Research, Denver, Colorado
  - Orhtopaedic Physicians Of Colorado, P.C., Englewood, Colorado
  - Orthopedics Assocs Of Hartford, Hartford, Connecticut
  - Anthony S. Unger, Md, Washington D.C., District of Columbia
  - Bay Pines Va Medical Center, Bay Pines, Florida
  - Pab Clinical Research, Brandon, Florida
  - Jacksonville Center For Clinical Research, Jacksonville, Florida
  - Mark W. Hollmann, Md, Orange City, Florida
  - Jewett Orthopaedic Clinic, Winter Park, Florida
  - Atlanta Knee And Sports Medicine, Decatur, Georgia
  - Americana Orthopedics, Boise, Idaho
  - Intermountain Orthopaedics, Boise, Idaho
  - Bluegrass Orthopaedics/Bmr, Lexington, Kentucky
  - Charleston Orthopaedic Assocs., Charleston, South Carolina
  - Kelsey Seybold Clinic, Houston, Texas
  - Bone & Joint Clinic Of Houston, Houston, Texas
  - Gill Orthopedic Center, Lubbock, Texas
  - Robert R. King, Md, Lubbock, Texas
  - Unlimited Research, San Antonio, Texas
- Argentina (3):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, Córdoba, Córdoba Province
- Australia (10):
  - Local Institution, Garran, Australian Capital Territory
  - Local Institution, Camperdown, New South Wales
  - Local Institution, Caringbah, New South Wales
  - Local Institution, Lismore, New South Wales
  - Local Institution, Gold Coast, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Bedford Park, South Australia
  - Local Institution, Box Hill, Victoria
  - Local Institution, Windsor, Victoria
  - Local Institution, Perth, Western Australia
- Brazil (5):
  - Local Institution, Curitiba, Paraná
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Porto Alegre, Rs, Rio Grande do Sul
  - Local Institution, Campinas, São Paulo
  - Local Institution, São Paulo, São Paulo
- Canada (19):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Ajax, Ontario
  - Local Institution, Burlington, Ontario
  - Local Institution, Cambridge, Ontario
  - Local Institution, Chatham, Ontario
  - Local Institution, Dartmouth, Ontario
  - Local Institution, Guelph, Ontario
  - Local Institution, Lindsay, Ontario
  - Local Institution, Newmarket, Ontario
  - Local Institution, Niagara Falls, Ontario
  - Local Institution, Sarnia, Ontario
  - Local Institution, Scarborough Village, Ontario
  - Local Institution, St. Catharines, Ontario
  - Local Institution, Stratford, Ontario
  - Local Institution, Waterloo, Ontario
  - Local Institution, Windsor, Ontario
  - Local Institution, Charlottetown, Prince Edward Island
  - Local Institution, Montreal, Quebec
  - Local Institution, Québec, Quebec
- Denmark (2):
  - Local Institution, Hørsholm
  - Local Institution, Kopenhamn S
- Hungary (3):
  - Local Institution, Kecskemét
  - Local Institution, Székesfehérvár
  - Local Institution, Szolnok
- Israel (8):
  - Local Institution, Afula
  - Local Institution, Beersheba
  - Local Institution, Haifa
  - Local Institution, Holon
  - Local Institution, Kfar Saba
  - Local Institution, Petah Tikva
  - Local Institution, Rehovot
  - Local Institution, Ẕerifin
- Mexico (8):
  - Local Institution, Chihuahua City, Chihuahua
  - Local Institution, Tijuana, Estado de Baja California
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Df, Mexico City
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Ciudad Madero, Tamaulipas
  - Local Institution, Jalapa, Veracruz
  - Local Institution, Mérida, Yucatán
- Poland (6):
  - Local Institution, Bialystok
  - Local Institution, Krakow
  - Local Institution, Lodz
  - Local Institution, Lublin
  - Local Institution, Szczecin
  - Local Institution, Warsaw
- Russia (3):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
  - Local Institution, Samara
- Local Institution, Gothenburg, Sweden
- Turkey (Türkiye) (4):
  - Local Institution, Adana
  - Local Institution, Bursa
  - Local Institution, Mersin
  - Local Institution, Trabzon

REFERENCES:
- [Derived] Jamieson MJ, Byon W, Dettloff RW, Crawford M, Gargalovic PS, Merali SJ, Onorato J, Quintero AJ, Russ C. Apixaban Use in Obese Patients: A Review of the Pharmacokinetic, Interventional, and Observational Study Data. Am J Cardiovasc Drugs. 2022 Nov;22(6):615-631. doi: 10.1007/s40256-022-00524-x. Epub 2022 May 16. PMID 35570249
- [Derived] Lassen MR, Raskob GE, Gallus A, Pineo G, Chen D, Portman RJ. Apixaban or enoxaparin for thromboprophylaxis after knee replacement. N Engl J Med. 2009 Aug 6;361(6):594-604. doi: 10.1056/NEJMoa0810773. PMID 19657123

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3608 patients enrolled and 3195 were randomized to double blind (DB) Treatment Period: 413 not randomized due to: 227 no longer met criteria, 109 withdrew consent, 60 other reasons, 11 administrative reason by sponsor, 5 adverse event, 1 poor, non-compliance.
Groups:
- Apixaban 2.5mg BID: Apixaban 2.5 mg tablets twice a day (BID) plus matching placebo SC injection q 12 hours for 12 days, plus or minus 2 days. The study included a screening period that began no more than 30 days prior to surgery through 24 hours after surgery; a 12 (±2) day treatment period, starting on the day of the first dose of study drug (day of surgery or next day); and a 60 (±3) day follow-up period, starting the day after the last dose of study drug (End of Treatment Period to Day 72).
- Enoxaparin 30 mg SC Injection q 12 Hours: Enoxaparin 30 mg subcutaneous (SC) injection every (q) 12 hours (h) plus matching placebo tablets BID for 12 days, plus or minus 2 days. The study included a screening period that began no more than 30 days prior to surgery through 24 hours after surgery; a 12 (±2) day treatment period, starting on the day of the first dose of study drug(day of surgery or next day); and a 60 (±3) day follow-up period, starting the day after the last dose of study drug (End of Treatment Period to Day 72).
Period: DB Treatment Period-Randomized Patients
Arm/Group | Apixaban 2.5mg BID | Enoxaparin 30 mg SC Injection q 12 Hours
Started | 1599 | 1596
Completed | 1509 | 1489
Not Completed | 90 | 107
Not completed — Death | 1 | 1
Not completed — Adverse Event | 60 | 58
Not completed — Withdrawal by Subject | 18 | 37
Not completed — Lost to Follow-up | 0 | 1
Not completed — No longer meets study criteria | 1 | 2
Not completed — Administrative reason by sponsor | 1 | 0
Not completed — non-specified | 9 | 8
Period: Follow-Up Period - Randomized Patients
Arm/Group | Apixaban 2.5mg BID | Enoxaparin 30 mg SC Injection q 12 Hours
Started | 1553 | 1533
Completed | 1492 | 1461
Not Completed | 61 | 72
Not completed — Withdrawal by Subject | 17 | 19
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 38 | 39
Not completed — non-specified | 6 | 12

BASELINE CHARACTERISTICS:
Population: Randomized participants were summarized.
Groups:
- Apixaban 2.5mg BID: Apixaban 2.5 mg tablets twice a day (BID) plus matching placebo SC injection q 12 hours for 12 days, plus or minus 2 days. The study included a screening period that began no more than 30 days prior to surgery through 24 hours after surgery; a 12 (±2) day treatment period, starting on the day of the first dose of study drug; and a 60 (±3) day follow-up period, starting the day after the last dose of study drug (End of Treatment Period to Day 72).
- Enoxaparin 30 mg SC Injection q 12 Hours: Enoxaparin 30 mg subcutaneous (SC) injection every (q) 12 hours (h) plus matching placebo tablets BID for 12 days, plus or minus 2 days. The study included a screening period that began no more than 30 days prior to surgery through 24 hours after surgery; a 12 (±2) day treatment period, starting on the day of the first dose of study drug; and a 60 (±3) day follow-up period, starting the day after the last dose of study drug (End of Treatment Period to Day 72).
- Total: Total of all reporting groups
Arm/Group | Apixaban 2.5mg BID | Enoxaparin 30 mg SC Injection q 12 Hours | Total
Number analyzed (Participants) | 1599 | 1596 | 3195
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (9.26) | 65.7 (9.22) | 65.8 (9.24)
Age, Customized [Number; unit: participants]
  Less than(<) 65 years | 697 | 691 | 1388
  Greater than, equal to (>=) 65 and < 75 years | 593 | 610 | 1203
  >=75 years | 309 | 295 | 604
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 997 | 986 | 1983
  Male | 602 | 610 | 1212
Region of Enrollment [Number; unit: participants]
  Argentina | 43 | 43 | 86
  Russian Federation | 15 | 13 | 28
  Hungary | 28 | 26 | 54
  United States | 464 | 474 | 938
  Canada | 554 | 548 | 1102
  Sweden | 66 | 68 | 134
  Turkey | 12 | 10 | 22
  Denmark | 87 | 89 | 176
  Brazil | 42 | 39 | 81
  Poland | 35 | 35 | 70
  Mexico | 138 | 138 | 276
  Israel | 44 | 42 | 86
  Australia | 50 | 54 | 104
  Norway | 21 | 17 | 38

OUTCOME MEASURES:

1. Primary Outcome: Event Rate of the Composite of Adjudicated Venous Thromboembolism (VTE) Events and All-Cause Death With Onset During the Intended Treatment Period - Primary Subjects
Description: An Independent Central Adjudication Committee (ICAC) adjudicated all venograms, suspected symptomatic deep vein thrombosis (DVT) and pulmonary embolism (PE), acute clinically overt bleeding events, suspected thrombocytopenia, suspected acute MI, suspected acute stroke, and cause of death. Event rate was number of participants with the composite endpoint divided by the number of participants analyzed and reported as percentage (%). Surgery=Day 1; Randomization/Treatment started on Day of Surgery or the next day (Day 1 or Day 2). A mandatory bilateral ascending contrast venogram was performed on all participants after 12 days (±2 days) of study treatment. Intended Treatment Period=starts on the day of randomization; for treated participants, the period ends at the latter of 2 days after last dose of study drug or 14 days after the first dose of study drug; for randomized participants who were not treated, the period ends 14 days after randomization.
Time Frame: From Day 1 or Day 2 to last dose, plus 2 days or 14 days post randomization
Population: Primary Population=All randomized participants who: have an adjudicated and evaluable bilateral venogram performed during the Intended Treatment Period; or have an adjudicated VTE during the Intended Treatment Period; or die due to any cause during the Intended Treatment Period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Apixaban 2.5mg BID: Apixaban 2.5 mg tablets twice a day (BID) plus matching placebo SC injection q 12 hours for 12 days, ± 2 days.
- Enoxaparin 30 mg SC Injection q 12 Hours: Enoxaparin 30 mg SC injection q 12 h plus matching placebo tablets BID for 12 days, ± 2 days.
Arm/Group | Apixaban 2.5mg BID | Enoxaparin 30 mg SC Injection q 12 Hours
Number analyzed (Participants) | 1157 | 1130
percentage of participants | 8.99 [7.47 to 10.79] | 8.85 [7.33 to 10.66]
Statistical Analysis 1: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Non-Inferiority or Equivalence — Two criteria were to be met to demonstrate non-inferiority: the upper bound of the 95% confidence interval (CI) for the Relative Risk should be < 1.25, and the upper bound of the 95% CI for the risk difference should be < 5.6%; p = 0.0635, t-test, 1 sided — If p-value is less than 0.025, it is statistically significant; Risk Ratio (RR) = 1.02, 95% CI 2-sided [0.78 to 1.32]
Statistical Analysis 2: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Non-Inferiority or Equivalence — Two criteria were to be met to demonstrate non-inferiority: the upper bound of the 95% CI for the relative risk should be < 1.25, and the upper bound of the 95% CI for the risk difference should be < 5.6%; p < 0.0001, t-test, 1 sided — If p-value is less than 0.025, it is statistically significant; Risk Difference (RD) = 0.11, 95% CI 2-sided [-2.22 to 2.44]

2. Secondary Outcome: Event Rate of Composite of Adjudicated Proximal DVT, Non-Fatal PE and All-Cause Death With Onset During the Intended Treatment Period PE and All-cause Death During the Intended Treatment Period
Description: A mandatory bilateral ascending contrast venogram was performed on all participants after 12 days (±2 days) of study treatment. An ICAC adjudicated all venograms, suspected proximal DVT and non-fatal PE, and all-cause of death. Event rate was number of participants with the composite endpoint divided by the number of participants analyzed and reported as percentage (%).
Time Frame: From Day 1 or Day 2 to last dose, plus 2 days or 14 days post randomization
Population: Randomized participants with either an adjudicated and evaluable bilateral proximal venogram or an adjudicated non-fatal PE or death, during the Intended Treatment Period, were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Apixaban 2.5mg BID: Apixaban 2.5 mg tablets BID plus matching placebo SC injection q 12 hours for 12 days, ±2 days.
- Enoxaparin 30 mg SC Injection q 12 Hours: Enoxaparin 30 mg SC injection q 12 hours plus placebo tablets BID for 12 days, ± 2 days.
Arm/Group | Apixaban 2.5mg BID | Enoxaparin 30 mg SC Injection q 12 Hours
Number analyzed (Participants) | 1269 | 1216
percentage of participants | 2.05 [1.39 to 3.01] | 1.64 [1.06 to 2.55]
Statistical Analysis 1: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Superiority or Other; Risk Ratio (RR) = 1.25, 95% CI 2-sided [0.70 to 2.23] — If the upper bound of the two-sided 95% CI for the Relative Risk was < 1 then superiority for the key secondary efficacy endpoint was demonstrated
Statistical Analysis 2: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Superiority or Other; Risk Difference (RD) = 0.36, 95% CI 2-sided [-0.68 to 1.40]
Statistical Analysis 3: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Superiority or Other; p = 0.7779, t-test, 1 sided

3. Secondary Outcome: Event Rate of Adjudicated VTE / VTE-related Death With Onset During the Treatment Period
Description: VTE / VTE-related death was defined as the combination of fatal or non-fatal PE, and symptomatic or asymptomatic DVT. A mandatory bilateral ascending contrast venogram was performed on all participants after 12 days (±2 days) of study treatment. An ICAC adjudicated all venograms, suspected symptomatic DVT and PE, and cause of death. Event rate was number of participants with the endpoint divided by the number of participant's analyzed (%).
Time Frame: From Day 1 or Day 2 to last dose, plus 2 days or 14 days post randomization
Population: Randomized participants with an adjudicated and evaluable bilateral venogram or an adjudicated event associated with the endpoint, during the Intended Treatment Period, were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Enoxaparin 30 mg SC Injection q 12 Hours: Enoxaparin 30 mg SC injection q 12 hours plus matching placebo tablets BID for 12 days, ±2 days.
Arm/Group | Apixaban 2.5mg BID | Enoxaparin 30 mg SC Injection q 12 Hours
Number analyzed (Participants) | 1156 | 1127
percentage of participants | 8.91 [7.40 to 10.71] | 8.61 [7.10 to 10.40]
Statistical Analysis 1: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Superiority or Other; Risk Ratio (RR) = 1.04, 95% CI 2-sided [0.80 to 1.35]
Statistical Analysis 2: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Superiority or Other; Risk Difference (RD) = 0.28, 95% CI 2-sided [-2.04 to 2.59]
Statistical Analysis 3: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Superiority or Other; p = 0.7754, test of equality — For descriptive purposes only, p-values were presented for the test of equality of event rates

4. Secondary Outcome: Event Rate for Participants With Proximal DVT/Non-Fatal PE/ VTE-Related Death With Onset During the Intended Treatment Period
Description: An ICAC adjudicated all venograms, suspected symptomatic DVT and PE, and cause of death. Event rate was number of participants with the endpoint divided by the number of participant's analyzed (%).
Time Frame: From Day 1 or Day 2 to last dose, plus 2 days or 14 days post randomization
Population: Randomized participants with either an adjudicated and evaluable bilateral proximal venogram or an adjudicated event associated with the endpoint, during the Intended Treatment Period, were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Enoxaparin 30 mg SC Injection q 12 Hours: Enoxaparin 30 mg SC injection q 12 hours plus matching placebo tablets BID for 12 days, ± 2 days.
Arm/Group | Apixaban 2.5mg BID | Enoxaparin 30 mg SC Injection q 12 Hours
Number analyzed (Participants) | 1268 | 1213
percentage of participants | 1.97 [1.33 to 2.92] | 1.40 [0.86 to 2.26]
Statistical Analysis 1: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Superiority or Other; Risk Ratio (RR) = 1.41, 95% CI 2-sided [0.77 to 2.60]
Statistical Analysis 2: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Superiority or Other; Risk Difference (RD) = 0.53, 95% CI 2-sided [-0.47 to 1.52]
Statistical Analysis 3: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Superiority or Other; p = 0.2626, test of equality — For descriptive purposes only, p-values were presented for the test of equality of event rates

5. Secondary Outcome: Event Rate for Total Participants With Adjudicated VTE/All-Cause Death With Onset During the Intended Treatment Period
Description: ICAC adjudicated all venograms, suspected symptomatic DVT and PE, and cause of death. Event rate was number of participants with the endpoint divided by the number of participant's analyzed (%).
Time Frame: From Day 1 or Day 2 to last dose, plus 2 days or 14 days post randomization
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apixaban 2.5mg BID | Enoxaparin 30 mg SC Injection q 12 Hours
Number analyzed (Participants) | 1270 | 1219
percentage of participants | 2.13 [1.46 to 3.10] | 1.97 [1.32 to 2.94]
Statistical Analysis 1: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Superiority or Other; Risk Ratio (RR) = 1.08, 95% CI 2-sided [0.63 to 1.87]
Statistical Analysis 2: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Superiority or Other; Risk Difference (RD) = 0.11, 95% CI 2-sided [-0.99 to 1.21]
Statistical Analysis 3: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Superiority or Other; p = 0.7700, test of equality — For descriptive purposes only, p-values were presented for the test of equality of event rates

6. Secondary Outcome: Event Rate for Total Participants With VTE/ VTE-Related Death With Onset During the Intended Treatment Period
Description: ICAC adjudicated all venograms, suspected symptomatic DVT and PE, and cause of death. VTE includes DVT and PE. Event rate was number of participants with the endpoint divided by the number of participant's analyzed (%).
Time Frame: From Day 1 or Day 2 to last dose, plus 2 days or 14 days post randomization
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apixaban 2.5mg BID | Enoxaparin 30 mg SC Injection q 12 Hours
Number analyzed (Participants) | 1269 | 1216
percentage of participants | 2.05 [1.39 to 3.01] | 1.73 [1.12 to 2.65]
Statistical Analysis 1: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Superiority or Other; Risk Ratio (RR) = 1.19, 95% CI 2-sided [0.68 to 2.11]
Statistical Analysis 2: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Superiority or Other; Risk Difference (RD) = 0.28, 95% CI 2-sided [-0.78 to 1.33]
Statistical Analysis 3: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Superiority or Other; p = 0.5443, test of equality; For descriptive purposes only, p-values were presented for the test of equality of event rates

7. Secondary Outcome: Event Rate for Participants With All-Cause Death During the Intended Treatment Period
Description: Event rate was number of participants with all-cause death divided by the number of participant's analyzed (%).
Time Frame: From Day 1 or Day 2 to last dose, plus 2 days or 14 days post randomization
Population: All Randomized participants were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apixaban 2.5mg BID | Enoxaparin 30 mg SC Injection q 12 Hours
Number analyzed (Participants) | 1599 | 1596
percentage of participants | 0.19 [0.04 to 0.59] | 0.19 [0.04 to 0.59]
Statistical Analysis 1: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Superiority or Other; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.20 to 4.93]
Statistical Analysis 2: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Superiority or Other; Risk Difference (RD) = 0.00, 95% CI 2-sided [-0.30 to 0.30]
Statistical Analysis 3: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Superiority or Other; p = 0.9975, test of equality — For descriptive purposes only, p-values were presented for the test of equality of event rates

8. Secondary Outcome: Event Rate for Participants With VTE-Related Death With Onset During the Intended Treatment Period
Description: ICAC adjudicated cause of death. Event rate was number of participants with the endpoint divided by the number of participant's analyzed (%).
Time Frame: From Day 1 or Day 2 to last dose, plus 2 days or 14 days post randomization
Population: All randomized participants were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Enoxaparin 30 mg SC Injection q 12 Hours: Enoxaparin 30 mg SC injection q 12 hours plus matching placebo tablets BID for 12 days,± 2 days.
Arm/Group | Apixaban 2.5mg BID | Enoxaparin 30 mg SC Injection q 12 Hours
Number analyzed (Participants) | 1599 | 1596
percentage of participants | 0.13 [0.00 to 0.49] | 0.00 [0.00 to 0.30]
Statistical Analysis 1: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Superiority or Other; Risk Difference (RD) = 0.13, 95% CI 2-sided [-0.05 to 0.30]
Statistical Analysis 2: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Superiority or Other; p = 0.1578, test of equality — For descriptive purposes only, p-values were presented for the test of equality of event rates

9. Secondary Outcome: Event Rate for Participants With Symptomatic VTE/ All-Cause Death With Onset During the Intended Treatment Period
Description: ICAC adjudicated suspected symptomatic DVT and PE, and cause of death. Event rate was number of participants with the endpoint divided by the number of participant's analyzed (%).
Time Frame: From Day 1 or Day 2 to last dose, plus 2 days or 14 days post randomization
Population: All randomized participants were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Apixaban 2.5mg BID: Apixaban 2.5 mg tablets BID) plus matching placebo SC injection q 12 hours for 12 days, ±2 days.
Arm/Group | Apixaban 2.5mg BID | Enoxaparin 30 mg SC Injection q 12 Hours
Number analyzed (Participants) | 1599 | 1596
percentage of participants | 1.25 [0.80 to 1.94] | 1.00 [0.61 to 1.64]
Statistical Analysis 1: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Superiority or Other; Risk Ratio (RR) = 1.25, 95% CI 2-sided [0.65 to 2.40]
Statistical Analysis 2: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Superiority or Other; Risk Difference (RD) = 0.25, 95% CI 2-sided [-0.47 to 0.98]

10. Secondary Outcome: Event Rate for Participants With Symptomatic VTE/ VTE-Related Death With Onset During the Intended Treatment Period
Description: as for outcome 9
Time Frame: From Day 1 or Day 2 to last dose, plus 2 days or 14 days post randomization
Population: All randomized participants were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apixaban 2.5mg BID | Enoxaparin 30 mg SC Injection q 12 Hours
Number analyzed (Participants) | 1599 | 1596
percentage of participants | 1.19 [0.75 to 1.87] | 0.81 [0.46 to 1.41]
Statistical Analysis 1: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Superiority or Other; Risk Ratio (RR) = 1.46, 95% CI 2-sided [0.72 to 2.95]
Statistical Analysis 2: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Superiority or Other; Risk Difference (RD) = 0.38, 95% CI 2-sided [-0.30 to 1.06]
Statistical Analysis 3: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Superiority or Other; p = 0.2873, test of equality — For descriptive purposes only, p-values were presented for the test of equality of event rates

11. Secondary Outcome: Event Rate for Participants With VTE/Major Bleeding/All-Cause Death With Onset During the Intended Treatment Period
Description: ICAC adjudicated VTE, acute clinically overt bleeding events, suspected thrombocytopenia, and cause of death. Event rate was number of participants with the composite endpoint divided by the number of participants analyzed (%).
Time Frame: From Day 1 or Day 2 to last dose, plus 2 days or 14 days post randomization
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apixaban 2.5mg BID | Enoxaparin 30 mg SC Injection q 12 Hours
Number analyzed (Participants) | 1162 | 1141
percentage of participants | 9.90 [8.31 to 11.76] | 10.60 [8.95 to 12.54]
Statistical Analysis 1: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Superiority or Other; Risk Ratio (RR) = 0.94, 95% CI 2-sided [0.74 to 1.20]
Statistical Analysis 2: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Superiority or Other; Risk Difference (RD) = -0.83, 95% CI 2-sided [-3.30 to 1.63]
Statistical Analysis 3: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Test type: Superiority or Other; p = 0.6145, test of equality — For descriptive purposes only, p-values were presented for the test of equality of event rates

12. Secondary Outcome: Event Rate for Participants With PE (Fatal or Non-Fatal), DVT (All, Symptomatic Proximal, and Distal, Asymptomatic) With Onset During the Intended Treatment Period
Description: An ICAC adjudicated all venograms, suspected symptomatic deep vein thrombosis (DVT) and pulmonary embolism (PE), acute clinically overt bleeding events, suspected thrombocytopenia, suspected acute MI, suspected acute stroke, and cause of death. Event rate was number of participants with the composite endpoint divided by the number of participants analyzed (%).
Time Frame: From Day 1 or Day 2 to last dose, plus 2 days or 14 days post randomization
Population: All randomized participants: PE, Symptomatic DVT, Symptomatic Proximal DVT, Symptomatic Distal DVT. Randomized with an adjudicated and evaluable bilateral venogram or an adjudicated event associated with the endpoint: All DVT, Asymptomatic DVT. n=number analyzed in each category
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apixaban 2.5mg BID | Enoxaparin 30 mg SC Injection q 12 Hours
Number analyzed (Participants) | 1599 | 1596
percentage of participants
  PE (Fatal or Non-Fatal) (n=1599, 1596) | 1.00 [0.61 to 1.64] | 0.44 [0.20 to 0.93]
  Non-Fatal PE (n=1599, 1596) | 0.88 [0.51 to 1.49] | 0.44 [0.20 to 0.93]
  All DVT n=1142, 1122 | 7.79 [6.37 to 9.51] | 8.20 [6.73 to 9.97]
  Symptomatic DVT (n=1599, 1596) | 0.19 [0.04 to 0.59] | 0.44 [0.20 to 0.93]
  Asymptomatic DVT (n=1139,1115) | 7.55 [6.15 to 9.25] | 7.62 [6.20 to 9.35]
  Symptomatic Proximal DVT (n=1599,1596) | 0.13 [0.00 to 0.49] | 0.19 [0.04 to 0.59]
  Symptomatic Distal DVT (n=1599,1596) | 0.06 [0.00 to 0.40] | 0.38 [0.15 to 0.85]

13. Secondary Outcome: Event Rate for Participants With Proximal DVT, Distal DVT, Asymptomatic Proximal DVT, Asymptomatic Distal DVT With Onset During the Intended Treatment Period
Description: ICAC adjudicated all venograms and suspected symptomatic DVT. Event rate was number of participants with the endpoint divided by the number of participant's analyzed (%).
Time Frame: From Day 1 or Day 2 to last dose, plus 2 days or 14 days post randomization
Population: Randomized participants with either an adjudicated and evaluable bilateral proximal (or distal, as appropriate) venogram or an adjudicated event associated with the endpoint. n= number analyzed
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apixaban 2.5mg BID | Enoxaparin 30 mg SC Injection q 12 Hours
Number analyzed (Participants) | 1254 | 1207
percentage of participants
  Proximal DVT (n=1254, 1207) | 0.72 [0.36 to 1.39] | 0.91 [0.49 to 1.65]
  Distal DVT (n=1146, 1133) | 7.24 [5.88 to 8.91] | 8.03 [6.58 to 9.78]
  Asymptomatic Proximal DVT (n=1252, 1204) | 0.56 [0.25 to 1.18] | 0.66 [0.32 to 1.34]
  Asymptomatic Distal DVT (n=1145, 1127) | 7.16 [5.80 to 8.82] | 7.54 [6.14 to 9.25]

14. Secondary Outcome: Event Rate for Participants With Adjudicated Myocardial Infarction (MI) Acute Ischemic Stroke and Thromboembolic Events With Onset During the Treatment Period
Description: ICAC adjudicated acute clinically overt bleeding events, suspected thrombocytopenia, suspected acute MI, suspected acute stroke per International Society on Thrombosis and Hemostasis (ISTH) guidelines modified for surgical patients. Event rate was number of participants with the composite endpoint divided by the number of participants analyzed (%).
Time Frame: From first dose to last dose, plus 2 days (12 days, plus 2)
Population: All participants who received at least one dose of study drug were analyzed (Treated Population).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apixaban 2.5mg BID | Enoxaparin 30 mg SC Injection q 12 Hours
Number analyzed (Participants) | 1596 | 1588
percentage of participants
  MI/Stroke | 0.06 [0.00 to 0.40] | 0.31 [0.11 to 0.77]
  MI | 0.06 [0.00 to 0.40] | 0.25 [0.08 to 0.68]
  Stroke | 0.00 [0.00 to 0.30] | 0.13 [0.01 to 0.50]
  Thrombocytopenia | 0.00 [0.00 to 0.30] | 0.13 [0.01 to 0.50]
Statistical Analysis 1: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Adjusted difference of event rates of MI/Stroke. Type of surgery was taken into consideration as a stratification factor; Test type: Superiority or Other; Risk Difference (RD) = -0.25, 95% CI 2-sided [-0.55 to 0.05]
Statistical Analysis 2: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Adjusted difference of event rates of MI. Type of surgery was taken into consideration as a stratification factor; Test type: Superiority or Other; Risk Difference (RD) = -0.19, 95% CI 2-sided [-0.46 to 0.09]
Statistical Analysis 3: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Adjusted difference of event rates of Stroke. Type of surgery was taken into consideration as a stratification factor; Test type: Superiority or Other; Risk Difference (RD) = -0.13, 95% CI 2-sided [-0.30 to 0.05]
Statistical Analysis 4: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Adjusted difference of event rates of thrombocytopenia. Type of surgery was taken into consideration as a stratification factor; Test type: Superiority or Other; Risk Difference (RD) = -0.13, 95% CI 2-sided [-0.30 to 0.05]

15. Primary Outcome: Event Rate for Participants With Major Bleeding, Clinically Relevant Non-Major Bleeding, Major or Clinically Relevant Non-Major Bleeding, Any Bleeding With Onset During the Treatment Period - Treated Population
Description: ICAC adjudicated acute clinically overt bleeding events as per International Society on Thrombosis and Hemostasis (ISTH) guidelines modified for surgical patients. Event rate was number of participants with the composite endpoint divided by the number of participants analyzed (%). Clinically relevant (CR); Non-Major (N-M) Bleeding. Day 1=Day of surgery. Treatment started (first dose) day of surgery or next day. Treatment continued for 12 days.
Time Frame: First dose of study drug to last dose, plus 2 days post last dose
Population: All participants who received at least one dose of study drug (Treated population).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Enoxaparin 30 mg SC Injection q 12 Hours: Enoxaparin 30 mg SC injection q 12 h plus matching placebo tablets BID for 12 days, ±2 days.
Arm/Group | Apixaban 2.5mg BID | Enoxaparin 30 mg SC Injection q 12 Hours
Number analyzed (Participants) | 1596 | 1588
percentage of participants
  Major Bleeding (n=1596, 1588) | 0.69 [0.37 to 1.25] | 1.39 [0.91 to 2.11]
  CR N-M Bleeding (n=1596, 1588) | 2.19 [1.58 to 3.05] | 2.96 [2.23 to 3.93]
  Major or CR N-M Bleeding(n=1596, 1588) | 2.88 [2.16 to 3.84] | 4.28 [3.39 to 5.41]
  Any Bleeding (n=1596, 1588) | 5.33 [4.33 to 6.55] | 6.80 [5.66 to 8.16]
Statistical Analysis 1: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Adjusted difference of event rates of Major Bleeding. Type of surgery was taken into consideration as a stratification factor; Test type: Superiority or Other; Risk Difference (RD) = -0.81, 95% CI 2-sided [-1.49 to -0.14]
Statistical Analysis 2: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Major Bleeding Endpoint; Test type: Superiority or Other; p = 0.0533, test of equality — For descriptive purposes only, p-values were presented for the test of equality of event rates
Statistical Analysis 3: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Adjusted difference of event rates of Clinically Relevant Non-Major Bleeding. Type of surgery was taken into consideration as a stratification factor; Test type: Superiority or Other; Risk Difference (RD) = -0.77, 95% CI 2-sided [-1.87 to 0.33]
Statistical Analysis 4: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Clinically relevant Non-Major Bleeding endpoint; Test type: Superiority or Other; p = 0.1709, test of equality — For descriptive purposes only, p-values were presented for the test of equality of event rates
Statistical Analysis 5: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Adjusted difference of event rates of Major or Clinically Relevant Non-Major Bleeding. Type of surgery was taken into consideration as a stratification factor; Test type: Superiority or Other; Risk Difference (RD) = -1.46, 95% CI 2-sided [-2.75 to -0.17]
Statistical Analysis 6: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Major or Clinically Relevant Non-Major Bleeding endpoint; Test type: Superiority or Other; p = 0.0338, test of equality; For descriptive purposes only, p-values were presented for the test of equality of event rates
Statistical Analysis 7: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Adjusted difference of event rates of Any Bleeding. Type of surgery was taken into consideration as a stratification factor; Test type: Superiority or Other; Risk Difference (RD) = -1.52, 95% CI 2-sided [-3.18 to 0.13]
Statistical Analysis 8: Comparison: Apixaban 2.5mg BID vs Enoxaparin 30 mg SC Injection q 12 Hours; Any Bleeding Endpoint; Test type: Superiority or Other; p = 0.0816, test of equality — For descriptive purposes only, p-values were presented for the test of equality of event rates

16. Primary Outcome: Event Rate for Participants With Major Bleeding, Clinically Relevant (CR) Non-Major (N-M) Bleeding , Major or Clinically Relevant (CR) Non-Major (N-M) Bleeding, Any Bleeding With Onset During the Follow-Up Period
Description: ICAC adjudicated acute clinically overt bleeding events as per International Society on Thrombosis and Hemostasis (ISTH) guidelines modified for surgical patients. Event rate was number of participants with the composite endpoint divided by the number of participants analyzed (%). Follow up Period was from the end of the treatment period (last dose) up to 60 days post last dose, Day 72.
Time Frame: Last dose of study drug to Day 72 (60 days)
Population: All participants who received at least 1 dose of study drug during the Treatment Period and entered the Follow-Up Period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Apixaban 2.5mg BID | Enoxaparin 30 mg SC Injection q 12 Hours
Number analyzed (Participants) | 1563 | 1553
percentage of participants
  Major Bleeding (n=1563, 1553) | 0.13 [0.01 to 0.51] | 0.13 [0.01 to 0.51]
  CR N-M Bleeding (n=1563, 1553) | 0.26 [0.08 to 0.69] | 0.45 [0.20 to 0.96]
  Major or CR N-M Bleeding (n=1563, 1553) | 0.38 [0.16 to 0.86] | 0.58 [0.29 to 1.12]
  Any Bleeding (n=1563, 1553) | 0.90 [0.52 to 1.52] | 1.29 [0.83 to 2.00]

17. Secondary Outcome: Event Rate of Adjudicated MI, Stroke, and Thrombocytopenia Events During the Follow-Up Period
Description: A 60-day follow-up period started after the last dose of study drug and continued until the End of Study Visit on Day 72 (60 days ± 3 days, after the last dose of study drug). Event rate was number of participants with the endpoint divided by the number of participants analyzed (%). ICAC adjudicated acute clinically overt bleeding events, suspected thrombocytopenia, suspected acute MI, suspected acute stroke per ISTH guidelines modified for surgical patients.
Time Frame: Post last dose of study drug to Day 72 (60 days)
Population: Participants who received at least one dose of study drug and entered the Follow-Up period
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Apixaban 2.5mg BID: Apixaban 2.5 mg tablets BID plus matching placebo SC injection q 12 hours for 12 days, plus or minus 2 days.
Arm/Group | Apixaban 2.5mg BID | Enoxaparin 30 mg SC Injection q 12 Hours
Number analyzed (Participants) | 1563 | 1553
percentage of participants
  MI/Stroke | 0.06 [0.00 to 0.41] | 0.06 [0.00 to 0.41]
  MI | 0.06 [0.00 to 0.41] | 0.06 [0.00 to 0.41]
  Stroke | 0.00 [0.00 to 0.30] | 0.00 [0.00 to 0.31]
  Thrombocytopenia | 0.00 [0.00 to 0.30] | 0.00 [0.00 to 0.31]

18. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Bleeding Adverse Events (AEs), AEs Leading to Discontinuation, and Deaths - Treated Population
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization.
Time Frame: First dose to last dose, plus 2 days for AEs (12 + 2 days) or plus 30 days for SAEs (12 + 30 days)
Population: All participants who received at least 1 dose of study drug during the Treatment Period.
Measure: Number; unit: participants
Groups:
- Enoxaparin 30 mg SC Injection q 12 Hours: Enoxaparin 30 mg SC injection q 12 h plus matching placebo tablets BID for 12 days, plus or minus 2 days.
Arm/Group | Apixaban 2.5mg BID | Enoxaparin 30 mg SC Injection q 12 Hours
Number analyzed (Participants) | 1596 | 1588
participants
  SAE | 123 | 123
  Bleeding AE | 110 | 144
  AEs leading to discontinuation | 60 | 58
  Deaths | 3 | 5

19. Secondary Outcome: Mean Change From Baseline in Systolic and Diastolic Blood Pressure During the Treatment Period
Description: Treatment Period=the period from first dose of study drug through 2 days after discontinuation of study drug (12 + 2 days). Baseline=measurement prior to first dose of study drug. Blood pressures (BP) were measured during screening (pre-operative, post-operative) and in the treatment period on Days 1 (day of first dose), 2, 3, 4,12 (end of treatment). Systolic and diastolic pressures were measured in millimeters of mercury (mmHg).
Time Frame: Baseline to last dose of study drug, plus 2 days
Population: All participants who received at least one dose of study drug and had blood pressure measurements at baseline were summarized.
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Apixaban 2.5mg BID | Enoxaparin 30 mg SC Injection q 12 Hours
Number analyzed (Participants) | 1577 | 1574
mmHg
  Diastolic BP Day 1 (n=240, 237) | -0.4 (0.741) | -0.9 (0.738)
  Diastolic BP Day 2 (n=1577, 1574) | 1.7 (0.301) | 1.5 (0.305)
  Diastolic BP Day 3 (n=1489,1498) | 2.3 (0.322) | 2.1 (0.321)
  Diastolic BP Day 4 (n=127,134) | 0.6 (1.217) | 0.3 (1.104)
  Diastolic BP Day 12 (n=1495,1463) | 7.3 (0.342) | 7.5 (0.343)
  Systolic BP Day 1 (n=240,237) | 1.5 (1.189) | -0.7 (1.303)
  Systolic BP Day 2 (n=1577,1574) | 5.4 (0.505) | 4.2 (0.518)
  Systolic BP Day 3 (n=1489,1498) | 4.7 (0.536) | 4.3 (0.555)
  Systolic BP Day 4 (n=127,134) | 2.8 (2.129) | 1.4 (1.871)
  Systolic BP Day 12 (n=1495,1463) | 9.1 (0.543) | 8.9 (0.562)

20. Secondary Outcome: Mean Change From Baseline in Heart Rate During the Treatment Period
Description: Treatment Period=the period from first dose of study drug through 2 days after discontinuation of study drug (12 + 2 days). Baseline=measurement prior to first dose of study drug. Heart rate was measured during screening (pre-operative, post-operative) and in the treatment period on Days 1 (day of first dose), 2, 3, 4,12 (end of treatment). Heart rate was measured in beats per minute (bpm).
Time Frame: Baseline to last dose of study drug, plus 2 days
Population: All participants who received at least one dose of study drug and had heart rate measurements at baseline were summarized.
Measure: Mean (Standard Error); unit: bpm
Arm/Group | Apixaban 2.5mg BID | Enoxaparin 30 mg SC Injection q 12 Hours
Number analyzed (Participants) | 1575 | 1574
bpm
  Heart Rate Day 1 (n=240,237) | 2.3 (0.761) | 2.7 (0.761)
  Heart Rate Day 2 (n=1575,1574) | 4.6 (0.312) | 4.5 (0.317)
  Heart Rate Day 3 (n=1490,1498) | 4.5 (0.334) | 5.0 (0.344)
  Heart Rate Day 4 (n=127,134) | 7.6 (1.365) | 9.4 (1.320)
  Heart Rate Day 12 (n=1495, 1462) | -0.3 (0.361) | -0.1 (0.375)

21. Secondary Outcome: Number of Participants With Hematology Laboratory Marked Abnormality During the Treatment Period
Description: Treatment Period=the period from first dose of study drug through 2 days after discontinuation of study drug. Hematology profile was measured during screening (pre-operative, post-operative) and in the Treatment Period on Days 2, 3, 4, 12 (end of treatment). Upper limit of normal (ULN); lower limit of normal (LLN). Platelet Count low: < 100,000/mm^3 (or < 100*109 cells/L). Erythrocytes low: < 0.75 *pre-dose. Hemoglobin low: > 2 g/dL decrease compared to pre-dose or Value ≤ 8 g/dL. Hematocrit low: < 0.75*pre-dose . Leukocytes: < 0.75*LLN or > 1.25* ULN, or if pre-dose < LLN then use < 0.8*predose or > ULN if pre-dose > ULN then use > 1.2*predose or < LLN. Lymphocytes (absolute): < 0.750*10^3 cells/µL or > 7.50*10^3 cells/ µL. Eosinophils (absolute) high: > 0.750*10^3 cells/µL. Basophils(absolute) high: > 400/mm^3 (or > 0.4*103 cells/µL). Monocytes (absolute) high: > 2000/mm^3 (or > 2*103 cells/µL). Neutrophils(absolute) high: < 1.0*103 cells/µL.
Time Frame: First dose to last dose of study drug (12 days), plus 2 days
Population: All participants who received at least one dose of study drug and had available laboratory results for that analyte and treatment group.
Measure: Number; unit: participants
Groups:
- Apixaban 2.5mg BID: Apixaban 2.5 mg tablets BID plus matching placebo SC injection q 12 hours for 12 days,± 2 days.
Arm/Group | Apixaban 2.5mg BID | Enoxaparin 30 mg SC Injection q 12 Hours
Number analyzed (Participants) | 1583 | 1572
participants
  Hemoglobin low (n=1561,1549) | 386 | 392
  Hematocrit low (n=1558,1547) | 135 | 157
  Platelet count low (n=1556,1543) | 6 | 9
  Erythrocytes low (n=1557,1547) | 130 | 149
  Leukocytes low(n=1583,1572) | 8 | 11
  Leukocytes high(n=1583,1572) | 214 | 210
  Basophils high (n=1577, 1564) | 0 | 2
  Eosinophils high (n=1577, 1564) | 32 | 13
  Lymphocytes low (n=1577,1564) | 125 | 117
  Lymphocytes high (n=1577,1564) | 2 | 4
  Monocytes high (n=1577,1564) | 4 | 4
  Neutrophils low (n=1577,1564) | 4 | 5

22. Secondary Outcome: Number of Participants With Liver and Kidney Function Chemistry Laboratory Marked Abnormalities During the Treatment Period
Description: Treatment Period=the period from first dose of study drug through 2 days after discontinuation of study drug. Laboratory Chemistry profile was measured during screening (pre-operative, post-operative) and in the Treatment Period on Days 4, and 12 (end of treatment). Bilirubin (direct) high: > 1.5*ULN. Total bilirubin: : > 2*ULN, Alanine Aminotransferase (ALT) high: > 3*ULN. Alkaline Phosphatase (ALP): > 2*ULN. Aspartate Aminotransferase (AST): > 3*ULN. Creatinine: > 1.5*ULN.
Time Frame: First dose to last dose of study drug (12 days), plus 2 days
Population: as for outcome 21
Measure: Number; unit: participants
Arm/Group | Apixaban 2.5mg BID | Enoxaparin 30 mg SC Injection q 12 Hours
Number analyzed (Participants) | 1573 | 1563
participants
  ALP high (n=1573,1563) | 42 | 55
  ALT high (n=1573,1562) | 33 | 45
  AST high (n=1573,1562) | 29 | 40
  Bilirubin direct high (n=1563,1553) | 63 | 54
  Bilirubin total high(n=1572,1562) | 2 | 8
  Creatinine high (n=1569,1562) | 17 | 28

23. Secondary Outcome: Number of Participants With Electrolyte Chemistry Laboratory Marked Abnormalities During the Treatment Period
Description: Laboratory Chemistry profile was measured during screening (pre-operative, post-operative) and in the Treatment Period on Days 4, and 12 (end of treatment). Potassium: < 0.9*LLN or > 1.1*ULN, or if pre-dose < LLN then use < 0.9*predose or > ULN if pre-dose > ULN then use > 1.1*predose or < LLN. Calcium: < 0.8*LLN or > 1.2*ULN, or if pre-dose < LLN then use < 0.75*predose or > ULN If pre-dose > ULN then use > 1.25*predose or < LLN. Chloride: < 0.9*LLN or > 1.1*ULN, or if pre-dose < LLN then use < 0.9*predose or > ULN if pre-dose > ULN then use > 1.1*predose or < LLN. Sodium: < 0.95*LLN or > 1.05*ULN, or if pre-dose < LLN then use < 0.95*predose or >ULN if pre-dose > ULN then use > 1.05*predose or < LLN. Bicarbonate: < 0.75*LLN or > 1.25*ULN, or if pre-dose < LLN then use < 0.75*predose or > ULN if pre-dose > ULN then use > 1.25*predose or < LLN.
Time Frame: First dose to last dose of study drug (12 days), plus 2 days
Population: as for outcome 21
Measure: Number; unit: participants
Arm/Group | Apixaban 2.5mg BID | Enoxaparin 30 mg SC Injection q 12 Hours
Number analyzed (Participants) | 1569 | 1562
participants
  Calcium low (n=1569,1562) | 1 | 5
  Calcium high (n=1569,1562) | 0 | 1
  Chloride low (n=1568,1562) | 11 | 17
  Chloride high (n=1568,1562) | 0 | 1
  Bicarbonate low (n=1568,1561) | 11 | 13
  Potassium low(n=1568,1559) | 54 | 56
  Potassium high(n=1568,1559) | 26 | 20
  Sodium low (n=1568,1562) | 23 | 39
  Sodium high (n=1568,1562) | 2 | 0

24. Secondary Outcome: Number of Participants With Other Chemistry Laboratory Marked Abnormalities During the Treatment Period
Description: Treatment Period=the period from first dose of study drug through 2 days after discontinuation of study drug. Laboratory Chemistry profile was measured during screening (pre-operative, post-operative) and in the Treatment Period on Days 4, and 12 (end of treatment). Fasting Glucose: if pre-dose < LLN then use < 0.8*predose; or > ULN if pre-dose > ULN then use > 2.0*predose or <LLN. Total Protein: < 0.9*LLN or > 1.1*ULN, or if pre-dose < LLN then use 0.9*predose or > ULN if pre-dose > ULN then use 1.1*predose or < LLN. Uric Acid: > 1.5*ULN, or if pre-dose > ULN then use > 2*predose. Creatine Kinase (CK): > 5*ULN.
Time Frame: First dose to last dose of study drug (12 days), plus 2 days
Population: as for outcome 21
Measure: Number; unit: participants
Arm/Group | Apixaban 2.5mg BID | Enoxaparin 30 mg SC Injection q 12 Hours
Number analyzed (Participants) | 1573 | 1563
participants
  Fasting Glucose low (n=611, 579) | 8 | 5
  Fasting Glucose high (n=611, 579) | 54 | 28
  Total Protein low (n=1568,1562) | 527 | 513
  CK high (n=1573,1563) | 52 | 45
  Uric Acid high (n=1567,1562) | 22 | 12

ADVERSE EVENTS:
Time Frame: First dose to last dose, plus 2 days for AEs or plus 30 days for SAEs.
Description: All participants who received at least one dose of study drug were included.
Arm/Group | Apixaban 2.5mg BID | Enoxaparin 30 mg SC Injection q 12 Hours
Serious Adverse Events (participants affected / at risk) | 123/1596 | 123/1588
Other Adverse Events (participants affected / at risk) | 713/1596 | 741/1588
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apixaban 2.5mg BID (N=1596) | Enoxaparin 30 mg SC Injection q 12 Hours (N=1588)
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 5 | 2
Atrial fibrillation (Cardiac disorders) | 3 | 5
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Hernia (General disorders) | 1 | 0
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Infection (Infections and infestations) | 2 | 0
Mania (Psychiatric disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 2
Pyelonephritis (Infections and infestations) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 1
Blood sodium decreased (Investigations) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 4
Chest discomfort (General disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0
Fat embolism (Injury, poisoning and procedural complications) | 1 | 0
Haematoma (Vascular disorders) | 3 | 4
Haemorrhage (Vascular disorders) | 0 | 2
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Heart rate increased (Investigations) | 1 | 0
Incision site infection (Infections and infestations) | 1 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Septic shock (Infections and infestations) | 1 | 0
Therapeutic response decreased (General disorders) | 0 | 1
Toxic encephalopathy (Nervous system disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 4 | 2
Wound secretion (Injury, poisoning and procedural complications) | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Blood pressure fluctuation (Vascular disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Cellulitis (Infections and infestations) | 4 | 2
Chest pain (General disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Gait disturbance (General disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 4
Oedema (General disorders) | 0 | 1
Post procedural infection (Infections and infestations) | 2 | 2
Skin infection (Infections and infestations) | 1 | 0
Syncope (Nervous system disorders) | 1 | 2
Vascular pseudoaneurysm (Vascular disorders) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 2
Bloody discharge (General disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Gastroenteritis (Infections and infestations) | 0 | 2
Heart rate decreased (Investigations) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Ileus (Gastrointestinal disorders) | 2 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 2
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Localised infection (Infections and infestations) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 2 | 2
Platelet count decreased (Investigations) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 2
Urinary retention (Renal and urinary disorders) | 1 | 1
Urosepsis (Infections and infestations) | 0 | 1
Wound haemorrhage (Vascular disorders) | 0 | 2
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 2
Calculus ureteric (Renal and urinary disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Clostridium difficile toxin test positive (Investigations) | 1 | 0
Delirium tremens (Psychiatric disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 5
Haemoglobin decreased (Investigations) | 1 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Incision site erythema (Injury, poisoning and procedural complications) | 1 | 0
Infusion site extravasation (General disorders) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Multi-organ failure (General disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1
Paronychia (Infections and infestations) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Blood culture positive (Investigations) | 0 | 1
Depression (Psychiatric disorders) | 0 | 2
Haematoma infection (Infections and infestations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Impaired healing (General disorders) | 0 | 2
Incision site pain (Injury, poisoning and procedural complications) | 1 | 0
Medical device complication (Injury, poisoning and procedural complications) | 1 | 1
Oxygen saturation decreased (Investigations) | 1 | 3
Postoperative wound infection (Infections and infestations) | 0 | 1
Secretion discharge (General disorders) | 1 | 1
Sedation (Nervous system disorders) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis infective (Infections and infestations) | 0 | 1
Asthenia (General disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Death (General disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 6 | 10
Encephalopathy (Nervous system disorders) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2
Joint contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Psychotic disorder (Psychiatric disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Swelling (General disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Bradycardia (Cardiac disorders) | 1 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 1
Discomfort (General disorders) | 1 | 0
Hypotension (Vascular disorders) | 2 | 1
Incision site cellulitis (Infections and infestations) | 1 | 1
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Oedema peripheral (General disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 2
Pneumonia (Infections and infestations) | 4 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Post procedural cellulitis (Infections and infestations) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 19 | 9
Pyrexia (General disorders) | 1 | 3
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 2 | 0
Weight decreased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Apixaban 2.5mg BID (N=1596) | Enoxaparin 30 mg SC Injection q 12 Hours (N=1588)
Vomiting (Gastrointestinal disorders) | 99 | 102
Insomnia (Psychiatric disorders) | 77 | 86
Dizziness (Nervous system disorders) | 103 | 88
Deep vein thrombosis (Vascular disorders) | 127 | 113
Nausea (Gastrointestinal disorders) | 208 | 241
Constipation (Gastrointestinal disorders) | 227 | 234
Oedema peripheral (General disorders) | 131 | 153
Pain in extremity (Musculoskeletal and connective tissue disorders) | 84 | 77
Pyrexia (General disorders) | 137 | 149

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.